CLINICAL TRIAL: NCT01480284
Title: A Multi-center, Randomized, Active Controlled, Double-blind, Parallel Group Comparison Study and Subsequent Open-label Study of GSK548470 in Patients With Compensated Chronic Hepatitis B Untreated With Nucleic Acid Analogue
Brief Title: Phase 3 Study of GSK548470 in Patients With Compensated Chronic Hepatitis B Untreated With Nucleic Acid Analogue
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 115409
Record Dates: First submitted 2011-11-23; First posted 2011-11-28 (Estimated); Results first posted 2013-10-29 (Estimated); Last update posted 2016-08-10 (Estimated); Status verified 2016-07

CONDITIONS: Hepatitis B, Chronic
Keywords: Tenofovir Disoproxil Fumarate; Chronic Hepatitis B
MeSH Terms: conditions — Hepatitis B, Chronic | interventions — Tablets; entecavir

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- GSK548470 300 mg (Experimental): GSK548470 300 mg tablet and ETV placebo capsule are administered once daily
  Interventions: Drug: GSK548470 300 mg tablet
- ETV 0.5 mg (Active Comparator): ETV 0.5 mg capsule and GSK548470 placebo tablet are administered once daily
  Interventions: Drug: ETV 0.5 mg capsule

INTERVENTIONS:
Drug: GSK548470 300 mg tablet — Blue tablets, each tablet containing 300 mg of tenofovir disoproxil fumarate
  Other Names: GSK548470
  Arms: GSK548470 300 mg
Drug: ETV 0.5 mg capsule — Brown capsules, each capsule containing 0.53 mg of entecavir hydrate
  Other Names: ETV
  Arms: ETV 0.5 mg

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of GSK548470 administered once daily at a dose level of 300 mg to Japanese patients with compensated chronic hepatitis B untreated with any nucleic acid analogue. In efficacy, the non-inferiority of GSK548470 to ETV will be verified using the antiviral effect as the index.

DETAILED DESCRIPTION:
This study is a multicenter, randomized, active comparator-controlled, double-blind, parallel-group comparison study in Japanese patients with compensated chronic hepatitis B untreated with any nucleic acid analogue and its subsequent open-label study. Efficacy and safety will be compared between once-daily dosing of GSK548470 300 mg and once-daily dosing of ETV 0.5 mg, and subsequently the efficacy and safety of GSK548470 administered long term will be investigated. A total of 165 subjects will be assigned to the GSK548470 group or the ETV group at a ratio of 2:1. The subjects will be assigned by stratified randomization in terms of HBe antigen and serum HBV-DNA level. The primary purpose is to verify the non-inferiority of GSK548470 to ETV using as an index the change amount of HBV-DNA level at Week 24 from the baseline level. The secondary purpose is to investigate the efficacy and safety of GSK548470 300 mg administered once daily for a long term.

ELIGIBILITY:
Inclusion Criteria:

* The ability to understand and sign a written informed consent form
* 16 to 69 years of age at the time of informed consent
* Females of childbearing potential must have a negative pregnancy test and agree to avoidance of pregnancy
* Subject must show QTc < 450 millisecond (msec) or < 480 msec with Bundle Branch Block
* Chronic HBV infection, defined as positive serum HBsAg for at least 6 month, or negative serum IgM-HBc antibody
* HBeAg positive; HBV-DNA >= 6 log10 copies/mL, HBeAg negative; HBV-DNA >= 5 log10 copies/mL
* Serum ALT >= 31 U/L and <= 10 × ULN
* Creatinine clearance >= 70 mL/min
* Haemoglobin >= 8 g/dL
* WBC >= 1,000 /mm3
* Nucleic acid analogue naïve, i.e., no prior therapy for over 6 months in the past
* No mutation that shows resistance in LAM, ETV and/or TDF at screening

Exclusion Criteria:

* Decompensated liver disease
* Co-infection with HIV or HCV
* Autoimmune hepatitis rather than chronic hepatitis B
* Subject with serious complication
* Received or have a plan for solid organ or bone marrow transplantation
* Has proximal tubulopathy
* History of hypersensitivity to nucleoside and/or nucleotide analogues
* Evidence of hepatocellular carcinoma by diagnostic imaging at screening and/or serum α-fetoprotein > 50 ng/mL at screening
* History of HCC
* Received any nucleoside, nucleotide, interferon or HB vaccine therapy within 24 weeks prior to initiation
* Received overdose NSAIDs, excluding temporary or topical use, within 7 days prior to initiation
* Received drugs for injection containing glycyrrhizin as the main component within 4 weeks prior to initiation
* Received drugs causing renal impairment, competitors of renal excretion, immunosuppressants, chemotherapeutics and/or corticosteroids within 8 weeks prior to initiation
* Participation in another clinical study within 6 months of study entry or planned participation in another clinical study after entry to this study
* Woman who is pregnant, lactating, possibly pregnant or planning a pregnancy during the study period
* Psychiatry disorder or cognitive disorder that may affect the subject ability to give informed consent or to follow specified study procedures
* History of alcohol or drug abuse
* Any condition or situation that may interfere with the subject's participation in the study

Ages: 16 Years to 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 166 (Actual)
Dates: Start 2011-11; Primary Completion 2013-01 (Actual); Study Completion 2014-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (19):
- Japan (19):
  - GSK Investigational Site, Aichi
  - GSK Investigational Site, Chiba
  - GSK Investigational Site, Fukui
  - GSK Investigational Site, Fukuoka
  - GSK Investigational Site, Gifu
  - GSK Investigational Site, Hiroshima
  - GSK Investigational Site, Hyōgo
  - GSK Investigational Site, Kagawa
  - GSK Investigational Site, Kagoshima
  - GSK Investigational Site, Kanagawa
  - GSK Investigational Site, Kumamoto
  - GSK Investigational Site, Miyagi
  - GSK Investigational Site, Miyazaki
  - GSK Investigational Site, Nagasaki
  - GSK Investigational Site, Nara
  - GSK Investigational Site, Okayama
  - GSK Investigational Site, Osaka
  - GSK Investigational Site, Saga
  - GSK Investigational Site, Tokyo

REFERENCES:
- [Derived] Koike K, Suyama K, Ito H, Itoh H, Sugiura W. Randomized prospective study showing the non-inferiority of tenofovir to entecavir in treatment-naive chronic hepatitis B patients. Hepatol Res. 2018 Jan;48(1):59-68. doi: 10.1111/hepr.12902. Epub 2017 May 24. PMID 28374496

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 166 participants (110 participants in the Tenofovir Disoproxil Fumarate [GSK548470, TDF] group and 56 participants in the Entecavir Hydrate [ETV] group) were enrolled in the study.
Groups:
- TDF 300 mg OD: Participants received Tenofovir Disoproxil Fumarate (TDF) 300 milligrams (mg) tablet once daily (OD) and Entecavir Hydrate (ETV) placebo capsule OD for 96 weeks.
- ETV 0.5 mg OD: Participants received ETV 0.5 mg capsule OD and TDF placebo tablet OD for 48 weeks.
Period: Overall Study
Arm/Group | TDF 300 mg OD | ETV 0.5 mg OD
Started | 110 | 56
Completed | 102 | 56
Not Completed | 8 | 0
Not completed — Withdrawal by Subject | 2 | 0
Not completed — Adverse Event | 1 | 0
Not completed — Study closed/terminated | 3 | 0
Not completed — Lost to Follow-up | 1 | 0
Not completed — Physician Decision | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- TDF 300 mg OD: Participants received TDF 300 mg tablet OD and ETV placebo capsule OD for 96 weeks.
- Total: Total of all reporting groups
Arm/Group | TDF 300 mg OD | ETV 0.5 mg OD | Total
Number analyzed (Participants) | 109 | 56 | 165
Age, Continuous [Mean (Standard Deviation); unit: Years] — Baseline characteristics are presented for the full analysis set, which is defined as all participants who entered into the study, received at least one dose of investigational product, and have at least one efficacy assessment after the treatment initiation.
  Years | 45.4 (9.23) | 46.1 (9.68) | 45.6 (9.36)
Sex: Female, Male [Count of Participants; unit: Participants] — Baseline characteristics are presented for the full analysis set, which is defined as all participants who entered into the study, received at least one dose of investigational product, and have at least one efficacy assessment after the treatment initiation.
  Participants
    Female | 41 | 16 | 57
    Male | 68 | 40 | 108
Race/Ethnicity, Customized [Number; unit: Participants] — Baseline characteristics are presented for the full analysis set, which is defined as all participants who entered into the study, received at least one dose of investigational product, and have at least one efficacy assessment after the treatment initiation.
  Participants
    Asian - Japanese Heritage | 109 | 56 | 165

OUTCOME MEASURES:

1. Primary Outcome: Mean Change From Baseline in Serum HBV DNA Level at Week 24
Description: The mean change from Baseline in the hepatitis B virus deoxyribonucleic acid (HBV DNA) level at Week 24 was assessed (lower limit of quantitation : 2.1 log 10 copies/mL). The mean values were adjusted by Baseline HBV DNA levels. Change from Baseline was calculated as the post-Baseline value minus the Baseline value.
Time Frame: Baseline and Week 24
Population: Per Protocol Set (PPS) Population: all participants who received at least 1 dose of investigational product (IP) and had at least one efficacy assessment after the treatment initiation, and with no major protocol violations. Missing values observed during the treatment period were imputed by the last observation carried forward (LOCF) method.
Measure: Least Squares Mean (Standard Error); unit: log10 copies/milliliter (copies/mL)
Arm/Group | TDF 300 mg OD | ETV 0.5 mg OD
Number analyzed (Participants) | 106 | 53
log10 copies/milliliter (copies/mL) | -4.63 (0.044) | -4.50 (0.063)
Statistical Analysis 1: Comparison: TDF 300 mg OD vs ETV 0.5 mg OD; Test type: Non-Inferiority or Equivalence — Non-inferiority was judged based on the one-sided test of the model, y(Δ) = Baseline + Group ( Δ= -1.0). The adjusted mean values of the TDF group and the ETV group were calculated, and the adjusted mean value and two-sided 95% confidence interval of differences between the TDF group and the ETV group were calculated. Non-inferiority was also to be confirmed when the upper limit of the calculated two-sided 95% confidence interval was less than the non-inferiority limit value of 1.0; p < 0.0001, ANCOVA — p-value was compared with the significance level of 0.025; Mean Difference (Final Values) = -0.13, 95% CI 2-sided [-0.28 to 0.02]

2. Secondary Outcome: Mean Change From Baseline in Serum HBV DNA Level at Week 48 and Week 96
Description: The mean change from Baseline in the HBV DNA level at Week 48 and Week 96 were assessed (lower limit of quantitation : 2.1 log10 copies/mL). The mean values were adjusted by Baseline HBV DNA levels. Change from Baseline was calculated as the post-baseline value minus the Baseline value. The LOCF method was applied for missing values.
Time Frame: Baseline, Week 48 and Week 96
Population: Full Analysis Set (FAS) Population: all participants who entered into the study, received at least one dose of investigational product, and have at least one efficacy assessment after the treatment initiation.
Measure: Mean (Standard Deviation); unit: log10 copies/mL
Arm/Group | TDF 300 mg OD | ETV 0.5 mg OD
Number analyzed (Participants) | 109 | 56
log10 copies/mL
  Week 48 | -4.86 (1.353) | -4.85 (0.916)
  Week 96 | -4.96 (1.445) | NA (NA) — Participants assigned to the arm ETV 0.5 mg OD completed the study at Week 48; therefore, there are no results for Week 96.
Statistical Analysis 1: Comparison: TDF 300 mg OD vs ETV 0.5 mg OD; Test type: Superiority or Other; Mean Difference (Final Values) = -0.01, 95% CI 2-sided [-0.40 to 0.39] — CI and estimate difference is provided for change from Baseline in serum HBV DNA level at Week 48

3. Secondary Outcome: Number of Participants With Serum HBV DNA < 2.1 log10 Copies/mL at Week 24, Week 48 and Week 96
Description: The number of participants with serum HBV DNA level less than the lower limit of quantitation (i.e. 2.1 log10 copies/mL) at Week 24, Week 48 and Week 96 were summarized. The LOCF method was applied for missing values.
Time Frame: Week 24, Week 48 and Week 96
Population: FAS Population
Measure: Number; unit: Participants
Arm/Group | TDF 300 mg OD | ETV 0.5 mg OD
Number analyzed (Participants) | 109 | 56
Participants
  Week 24 | 59 | 22
  Week 48 | 84 | 37
  Week 96 | 97 | NA — Participants assigned to the arm ETV 0.5 mg OD completed the study at Week 48; therefore, there are no results for Week 96.

4. Secondary Outcome: Number of Participants With Alanine Aminotransferase (ALT) Normalization at Week 24, Week 48 and Week 96
Description: The number of participants with alanine aminotransferase (ALT) normalization at Week 24, Week 48 and Week 96 were summarized. ALT normalization is defined as when an ALT value exceeds the upper limit of normal range (ULN) at Baseline and within the normal range at the end of treatment. The LOCF method was applied for missing values.
Time Frame: Week 24, Week 48 and Week 96
Population: Biochemically Evaluable Population (BEP): all participants who received at least one dose of IP and with an abnormal ALT at Baseline. The population for the analysis of ALT normalization was all participants with an ALT value > ULN at Baseline.
Measure: Number; unit: Participants
Arm/Group | TDF 300 mg OD | ETV 0.5 mg OD
Number analyzed (Participants) | 83 | 41
Participants
  Week 24 | 58 | 35
  Week 48 | 62 | 35
  Week 96 | 74 | NA — Participants assigned to the arm ETV 0.5 mg OD completed the study at Week 48; therefore, there are no results for Week 96.

5. Secondary Outcome: Number of Participants With HBeAg Loss at Week 24, Week 48 and Week 96
Description: The number of participants achieving hepatitis Be antigen (HBeAg) loss at Week 24, Week 48 and Week 96 in positive HBeAg participants at Baseline were summarized. Loss of HBeAg is defined as the change of detectable HBeAg from positive to negative. The LOCF method was applied for missing values.
Time Frame: Week 24, Week 48 and Week 96
Population: FAS Population. Only participants with positive HBeAg at Baseline were analyzed.
Measure: Number; unit: Participants
Arm/Group | TDF 300 mg OD | ETV 0.5 mg OD
Number analyzed (Participants) | 51 | 28
Participants
  Week 24 | 3 | 2
  Week 48 | 9 | 3
  Week 96 | 13 | NA — Participants assigned to the arm ETV 0.5 mg OD completed the study at Week 48; therefore, there are no results for Week 96.

6. Secondary Outcome: Number of Participants With HBeAg/HBeAb Seroconversion at Week 24, Week 48 and Week 96
Description: The number of participants achieving HBeAg/hepatitis Be antibody (HBeAb) seroconversion at Week 24, Week 48 and Week 96 in positive HBeAg and negative HBeAb participants at Baseline were summarized. Seroconversion to HBeAg is defined as the change of detectable antibody to HBeAg from negative to positive. The LOCF method was applied for missing values.
Time Frame: Week 24, Week 48 and Week 96
Population: FAS Population. Only participants with positive HBeAg and negative HBeAb at Baseline were analyzed.
Measure: Number; unit: Participants
Arm/Group | TDF 300 mg OD | ETV 0.5 mg OD
Number analyzed (Participants) | 43 | 27
Participants
  Week 24 | 0 | 1
  Week 48 | 4 | 2
  Week 96 | 5 | NA — Participants assigned to the arm ETV 0.5 mg OD completed the study at Week 48; therefore, there are no results for Week 96.

7. Secondary Outcome: Number of Participants Achieving HBsAg Loss at Week 24, Week 48 and Week 96
Description: The number of participants with hepatitis B surface antigen (HBsAg) loss at Week 24, Week 48 and Week 96 in positive HBsAg participants at Baseline were summarized. Loss of HBsAg is defined as change of detectable HBsAg from positive to negative. The LOCF method was applied for missing values.
Time Frame: Week 24, Week 48 and Week 96
Population: FAS Population.
Measure: Number; unit: Participants
Arm/Group | TDF 300 mg OD | ETV 0.5 mg OD
Number analyzed (Participants) | 109 | 56
Participants
  Week 24 | 0 | 0
  Week 48 | 0 | 0
  Week 96 | 1 | NA — Participants assigned to the arm ETV 0.5 mg OD completed the study at Week 48; therefore, there are no results for Week 96.

8. Secondary Outcome: Number of Participants Achieving HBsAg/HBsAb Seroconversion at Week 24, Week 48 and Week 96
Description: The number of participants with HBsAg/hepatitis B surface antibody (HBsAb) seroconversion at Week 24, Week 48 and Week 96 in positive HBsAg and negative HBsAb participants at Baseline were summarized. HBsAg seroconversion .is defined as change of detectable antibody to HBsAg from negative to positive. The LOCF method was applied for missing values.
Time Frame: Week 24, Week 48 and Week 96
Population: FAS Population. Only participants with positive HBsAg and negative HBsAb at Baseline were analyzed.
Measure: Number; unit: Participants
Arm/Group | TDF 300 mg OD | ETV 0.5 mg OD
Number analyzed (Participants) | 104 | 53
Participants
  Week 24 | 0 | 0
  Week 48 | 0 | 0
  Week 96 | 1 | NA — Participants assigned to the arm ETV 0.5 mg OD completed the study at Week 48; therefore, there are no results for Week 96.

9. Secondary Outcome: Number of Participants Achieving Each Indicated HBsAg Category at Baseline, Week 24, Week 48 and Week 96
Description: The number of participants achieving each indicated HBsAg category (HBsAg <80, 80 to 800, 800 to 8000, 8000 to 80000, and >=80000) (kilo international unit per liter [KIU/L]) by study visit was summarized. The LOCF method was applied for missing values.
Time Frame: Baseline, Week 24, Week 48 and Week 96
Population: FAS Population
Measure: Number; unit: Participants
Arm/Group | TDF 300 mg OD | ETV 0.5 mg OD
Number analyzed (Participants) | 109 | 56
Participants
  HBsAg <80 KIU/L, Baseline | 2 | 2
  HBsAg 80-800 KIU/L, Baseline | 15 | 10
  HBsAg 800-8000 KIU/L, Baseline | 58 | 33
  HBsAg 8000-80,000 KIU/L, Baseline | 31 | 10
  HBsAg >=80,000 KIU/L, Baseline | 3 | 1
  HBsAg <80 KIU/L, Week 24 | 3 | 1
  HBsAg 80-800 KIU/L, Week 24 | 17 | 10
  HBsAg 800-8000 KIU/L, Week 24 | 63 | 36
  HBsAg 8000-80,000 KIU/L, Week 24 | 26 | 9
  HBsAg >=80,000 KIU/L, Week 24 | 0 | 0
  HBsAg <80 KIU/L, Week 48 | 5 | 1
  HBsAg 80-800 KIU/L, Week 48 | 19 | 9
  HBsAg 800-8000 KIU/L, Week 48 | 60 | 39
  HBsAg 8000-80,000 KIU/L, Week 48 | 25 | 7
  HBsAg >=80,000 KIU/L, Week 48 | 0 | 0
  HBsAg <80 KIU/L, Week 96 | 5 | NA — Participants assigned to the arm ETV 0.5 mg OD completed the study at Week 48; therefore, there are no results for Week 96.
  HBsAg 80-800 KIU/L, Week 96 | 23 | NA — Participants assigned to the arm ETV 0.5 mg OD completed the study at Week 48; therefore, there are no results for Week 96.
  HBsAg 800-8000 KIU/L, Week 96 | 60 | NA — Participants assigned to the arm ETV 0.5 mg OD completed the study at Week 48; therefore, there are no results for Week 96.
  HBsAg 8000-80,000 KIU/L, Week 96 | 21 | NA — Participants assigned to the arm ETV 0.5 mg OD completed the study at Week 48; therefore, there are no results for Week 96.
  HBsAg >=80,000 KIU/L, Week 96 | 0 | NA — Participants assigned to the arm ETV 0.5 mg OD completed the study at Week 48; therefore, there are no results for Week 96.

10. Secondary Outcome: Number of Participants Achieving Each Indicated HBcrAg Category at Baseline, Week 24, Week 48 and Week 96
Description: The number of participants achieving each indicated hepatitis B core-related antigen (HBcrAg) category (HBcrAg <3.0, 3.0 to 4.0, 4.0 to 5.0, 5.0 to 6.0, and >=6.0) (Log kilo unit per liter [KU/L]) by study visit was summarized. The LOCF method was applied for missing values.
Time Frame: Baseline, Week 24, Week 48 and Week 96
Population: FAS Population
Measure: Number; unit: Participants
Arm/Group | TDF 300 mg OD | ETV 0.5 mg OD
Number analyzed (Participants) | 109 | 56
Participants
  HBcrAg <3.0 Log KU/L, Baseline | 7 | 0
  HBcrAg 3.0-4.0 Log KU/L, Baseline | 13 | 6
  HBcrAg 4.0-5.0 Log KU/L, Baseline | 19 | 11
  HBcrAg 5.0-6.0 Log KU/L, Baseline | 19 | 9
  HBcrAg >=6.0 Log KU/L, Baseline | 51 | 30
  HBcrAg <3.0 Log KU/L, Week 24 | 21 | 10
  HBcrAg 3.0-4.0 Log KU/L, Week 24 | 16 | 8
  HBcrAg 4.0-5.0 Log KU/L, Week 24 | 18 | 8
  HBcrAg 5.0-6.0 Log KU/L, Week 24 | 17 | 7
  HBcrAg >=6.0 Log KU/L, Week 24 | 37 | 23
  HBcrAg <3.0 Log KU/L, Week 48 | 24 | 12
  HBcrAg 3.0-4.0 Log KU/L, Week 48 | 16 | 6
  HBcrAg 4.0-5.0 Log KU/L, Week 48 | 18 | 9
  HBcrAg 5.0-6.0 Log KU/L, Week 48 | 23 | 10
  HBcrAg >=6.0 Log KU/L, Week 48 | 28 | 19
  HBcrAg <3.0 Log KU/L, Week 96 | 24 | NA — Participants assigned to the arm ETV 0.5 mg OD completed the study at Week 48; therefore, there are no results for Week 96.
  HBcrAg 3.0-4.0 Log KU/L, Week 96 | 18 | NA — Participants assigned to the arm ETV 0.5 mg OD completed the study at Week 48; therefore, there are no results for Week 96.
  HBcrAg 4.0-5.0 Log KU/L, Week 96 | 22 | NA — Participants assigned to the arm ETV 0.5 mg OD completed the study at Week 48; therefore, there are no results for Week 96.
  HBcrAg 5.0-6.0 Log KU/L, Week 96 | 23 | NA — Participants assigned to the arm ETV 0.5 mg OD completed the study at Week 48; therefore, there are no results for Week 96.
  HBcrAg >=6.0 Log KU/L, Week 96 | 22 | NA — Participants assigned to the arm ETV 0.5 mg OD completed the study at Week 48; therefore, there are no results for Week 96.

11. Secondary Outcome: Number of Participants With Virological Breakthrough Through End of the Study
Description: The number of participants who experienced virological breakthrough was summarized. Virological breakthrough is defined as serum HBV DNA level increase >=1 log10 copies/mL above the treatment nadir. Virological breakthrough values were presented from Baseline to through out the study. Baseline is defined as the value at Week 0 visit.
Time Frame: From Baseline to throughout study
Population: FAS Population
Measure: Number; unit: Participants
Arm/Group | TDF 300 mg OD | ETV 0.5 mg OD
Number analyzed (Participants) | 109 | 56
Participants | 2 | 2

12. Secondary Outcome: Number of Participants With Resistance Related Mutations at Week 24, Week 48, Week 96 and Virological Breakthrough (Baseline to Throughout the Study)
Description: The development of drug resistance-related (RA) mutations was analyzed to look for resistance to Lamivudine (LAM), Adefovir dipivoxil (ADV), and/or ETV in a case where a virologic breakthrough has been observed after starting the study treatment (serum HBV DNA level has increased from the nadir by at least 1 log10 copies/mL) or where the serum HBV DNA level is not less than the HBV DNA detection limit (2.1 log10 copies/mL) at Week 24, Week 48 and Week 96. Virologic breakthrough was defined as 1.0 log10 or greater increases in serum HBV-DNA levels from on-treatment nadir. Participants who achieved the HBV-DNA values below lower limit of quantification (LLQ) (< 2.1 log10 copies/mL) in quantitative analysis at entire the study were also considered "Negative" in drug-resistance without implementation of genotypic analysis. Resistance mutation values were presented from Baseline to throughout the study. Baseline is defined as the value at Week 0 visit.
Time Frame: Screening, Week 24, Week 48, Week 96 and Virological Breakthrough (Baseline to throughout the study)
Population: FAS Population. Only those participants available at the specified time points were analyzed (represented by n=X, X in the category titles).
Measure: Number; unit: Participants
Arm/Group | TDF 300 mg OD | ETV 0.5 mg OD
Number analyzed (Participants) | 109 | 56
Participants
  LAM RA mutations, Screening, n=109, 56 | 0 | 0
  ADV RA mutations, Screening, n=109, 56 | 0 | 0
  ETV RA mutations, Screening, n=109, 56 | 0 | 0
  LAM RA mutations, Week 24, n=49, 34 | 0 | 0
  ADV RA mutations, Week 24, n=49, 34 | 0 | 0
  ETV RA mutations, Week 24, n=49, 34 | 0 | 0
  LAM RA mutations, Week 48, n=23, 19 | 0 | 0
  ADV RA mutations, Week 48, n=23, 19 | 0 | 0
  ETV RA mutations, Week 48, n=23, 19 | 0 | 0
  LAM RA mutations, Week 96, n=11, 0 | 0 | NA — Participants assigned to the arm ETV 0.5 mg OD completed the study at Week 48; therefore, there are no results for Week 96.
  ADV RA mutations, Week 96, n=11, 0 | 0 | NA — Participants assigned to the arm ETV 0.5 mg OD completed the study at Week 48; therefore, there are no results for Week 96.
  ETV RA mutations, Week 96, n=11, 0 | 0 | NA — Participants assigned to the arm ETV 0.5 mg OD completed the study at Week 48; therefore, there are no results for Week 96.
  LAM RA mutations, Virologic Breakthrough, n=2, 2 | 0 | 0
  ADV RA mutations, Virologic Breakthrough, n=2, 2 | 0 | 0
  ETV RA mutations, Virologic Breakthrough, n=2, 2 | 0 | 0

ADVERSE EVENTS:
Time Frame: Serious adverse events (SAEs) and non-serious AEs were collected from the start of study medication to the end of the treatment period (up to average of 96 weeks).
Description: SAEs and non-serious AEs were collected in members of the Safety Population, comprised of all participants who received at least one dose of investigational product.
Arm/Group | TDF 300 mg OD | ETV 0.5 mg OD
Serious Adverse Events (participants affected / at risk) | 7/109 | 2/56
Other Adverse Events (participants affected / at risk) | 83/109 | 40/56
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | TDF 300 mg OD (N=109) | ETV 0.5 mg OD (N=56)
Arrhythmia (Cardiac disorders) | 1 | 0
Food poisoning (Gastrointestinal disorders) | 1 | 0
Urinary tract infection (Infections and infestations) | 1 | 0
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 2 | 0
Large intestine polyp (Gastrointestinal disorders) | 0 | 1
Dizziness (Nervous system disorders) | 1 | 0
Multiple fractures (Injury, poisoning and procedural complications) | 1 | 0
Hepatocellular carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Ovarian germ cell teratoma benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | TDF 300 mg OD (N=109) | ETV 0.5 mg OD (N=56)
Nasopharyngitis (Infections and infestations) | 48 | 24
Headache (Nervous system disorders) | 16 | 5
Blood creatine phosphokinase increased (Investigations) | 11 | 4
Influenza (Infections and infestations) | 10 | 3
Pharyngitis (Infections and infestations) | 10 | 2
Sinusitis (Infections and infestations) | 7 | 3
Oral herpes (Infections and infestations) | 6 | 0
Dizziness (Nervous system disorders) | 6 | 2
Lipase increased (Investigations) | 6 | 2
Abdominal pain upper (Gastrointestinal disorders) | 8 | 0
Dental caries (Gastrointestinal disorders) | 4 | 4
Diarrhoea (Gastrointestinal disorders) | 5 | 3
Constipation (Gastrointestinal disorders) | 3 | 3
Back pain (Musculoskeletal and connective tissue disorders) | 6 | 4
Myalgia (Musculoskeletal and connective tissue disorders) | 4 | 3
Cough (Respiratory, thoracic and mediastinal disorders) | 7 | 2
Rash (Skin and subcutaneous tissue disorders) | 2 | 5
Seasonal allergy (Immune system disorders) | 1 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.